CLINICAL TRIAL: NCT06802341
Title: Energy Metabolism and Acute Effects of Protein Diets in Metabolically Obese Normal Weight (MONW) Individuals
Brief Title: Energy Metabolism and Acute Effects of Protein Diets in Metabolically Obese Normal Weight Individuals
Acronym: MONW
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Responsible Party: Principal Investigator, Melvin Leow, Prof Melvin Leow Khee-Shing, Singapore Institute of Food and Biotechnology Innovation
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2021-192
Record Dates: First submitted 2025-01-17; First posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Healthy; Glucose Metabolism Disorders; Obesity, Visceral; Obesity; Endocrine; Insulin Sensitivity; Insulin Resistance
Keywords: Glycaemic control
MeSH Terms: conditions — Glucose Metabolism Disorders; Obesity, Abdominal; Obesity; Insulin Resistance | interventions — Diet, Plant-Based

STUDY DESIGN:
Intervention Model Description: Randomized, controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Normal protein diet (Experimental): Animal based protein. 60% carbohydrates, 10% proteins and 30% lipids (i.e. 0.8g of protein/kg of body weight/day)
  Interventions: Other: Normal protein diet
- Animal based high protein meal (Experimental): 40% carbohydrates, 30% proteins and 30% lipids (i.e. 2.4g of protein/kg of body weight/day)
  Interventions: Other: Animal protein diet
- Plant based high protein meal (Experimental): 40% carbohydrates, 30% proteins and 30% lipids (i.e. 2.4g of protein/kg of body weight/day)
  Interventions: Other: Plant based diet

INTERVENTIONS:
Other: Normal protein diet — Animal-based protein meal plan consisted of 60% carbohydrates, 10% proteins and 30% lipids
  Arms: Normal protein diet
Other: Animal protein diet — Animal based high protein meal consisting of 40% carbohydrates, 30% proteins and 30% lipids
  Arms: Animal based high protein meal
Other: Plant based diet — Plant based high protein meal consisting of 40% carbohydrates, 30% proteins and 30% lipids
  Arms: Plant based high protein meal

SUMMARY:
Asians tend to develop type 2 diabetes (T2D) at lower body mass index (BMI) levels and younger ages compared to other populations. This leads to a longer duration of suffering from long-term complications associated with the disease, ultimately resulting in shorter life expectancy. Notably, approximately 40% of newly diagnosed T2D cases in Asians occur in individuals considered lean, with a BMI reported to be less than 22 kg/m2. This phenomenon is termed the "Metabolically Obese Normal Weight" (MONW) phenotype. MONW individuals are characterized as having a normal body weight but exhibiting obesity-related metabolic disturbances, including excess body fat with ectopic fat deposition, insulin resistance, and dyslipidemia.

DETAILED DESCRIPTION:
Asian populations have higher prevalence of abdominal obesity, accounting for ~60% of the global diabetic population. Type 2 diabetes (T2D) developing at lower BMI levels and younger ages compared to Western populations, suggest underlying metabolic issues in Asian. A cluster of metabolically obese, normal weight (MONW) individuals are identified in 40% of newly diagnosed Asian T2D.

MONW individuals have normal body weight but exhibit obesity-related metabolic disturbances, such as excess body fat, insulin resistance, and dyslipidemia, predisposing them to develop metabolic symptoms such as T2D and cardiovascular disease. They also show reduced physical activity, lower aerobic capacity, low muscle quality and impaired thermogenesis. Elevated plasma amino acids are associated with insulin resistance, resembling obesity, diabetes and sarcopenia. Given the complex nature of MONW, further examination is needed for early diagnosis and effective prevention strategies. Increased protein intake is known to improve satiety, thermogenesis and muscle health, while enhancing insulin sensitivity and fat oxidation. High-protein diets can aid in weight loss and are often preferred over traditional calorie restriction for combating obesity. In our previous study, a 5% weight loss from calorie restriction improved body composition and metabolism in MONW individuals. Hence, this study aims to 1) better understand the physiology and energy balance of MONW individuals; 2) identify biomarkers for early diagnosis; and 3) examine the effects of high-protein diets on the metabolism of MONW individuals. The study will involve participants of Chinese descent, evaluating metabolic biomarkers in energy balance and the impact of different protein sources on their acute metabolic effects.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between 18.5 - 24.9 kg/m2
* Non-diabetic
* Blood pressure (≤140/90 mmHg)
* <5% weight change in the past 6 months
* Fasting triglyceride < 90 mg/dl and HOMA-IR ≤ 1.0 will be defined as healthy subjects
* Fasting triglyceride ≥ 90 mg/dl and HOMA-IR > 1.0 will be defined as MONW subjects

Exclusion Criteria:

* • Smoker or currently on nicotine therapy

  * Regularly consume alcohol >1 unit per day
  * On hypocaloric/hypercaloric diet aiming for weight loss/gain
  * An athlete or sportive person with regular exercising >3 times per week and >45 minutes per section.
  * Currently receiving therapy (e.g. insulin) or any medication/ treatment (including supplements) that may affect glucose and lipid metabolism, energy metabolism or body composition
  * Currently on steroids, protease inhibitors, or antipsychotics therapies
  * Has symptomatic Irritable Bowel Syndrome
  * Has glucose-6-phosphate dehydrogenase (G6PD) deficiency
  * Had major medical or surgical event requiring hospitalization within the preceding 3 months
  * Participated in drug trials within 3 months before the start of the study
  * Donated blood within 3 months before the start of the study
  * Has intolerances or allergies to any of the study foods (eg. anaphylaxis to glutens)
  * Pregnant (pregnancy test will be done), lactating, or planning to be become pregnant during the study period
  * Has active Tuberculosis (TB) or currently receiving treatment for TB
  * Has chronic infection or is known to suffer from or has previously suffered from or is a carrier of Hepatitis B Virus (HBV), Hepatitis C Virus (HCV), Human Immunodeficiency Virus (HIV)
  * Has claustrophobia, trypanophobia, or hemophobia
  * Unwilling to consume study foods
  * Inadequate fluency in the English language
  * Unable to understand the study procedures and signs forms providing written informed consent to participate in the study.
  * Is a member of the research team or their immediate family members. Immediate family member is defined as a spouse, parent, child, or sibling, whether biological or legally adopted

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Males and females
Enrollment: 24 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Gycaemic control | Blood will be sampled at timepoints, t = 0minute(fasting), following the meal test,for 4 hours (t = 15, 30, 60, 90, 120, 150, 180 and 240 minutes),and pre- and post-exercise
  The primary outcome in this study is the effect on glycaemic control (fasting glucose, insulin, insulin sensitivity).
Energy expenditure and fuel utilization | Assessed for 9 hours in the whole body calorimeter room on visits 3, 4 and 5. 30 minute-RMR,3hour-DIT, 30minute-exercise-induced EE (or PAEE)); urine samples collected on 4 different sessions throughout the WBC
  Metabolism will be assessed in the whole body calorimeter (WBC). Only one subject alone in the WBC room during the test. The subject can move around freely. O2 consumption and CO2 production will be detailed energy metabolism in different parameters, such as RMR, DIT, PAEE and NEAT.measured to calculate energy expenditure using Weir formulae Urine samples collected across 4 different sessions throughout the WBC stay to assess protein utilisation
Postprandial amino acids and proteomics profiles | Blood will be sampled at timepoints, t = 0 minute (Baseline) and at t=60 minutes.
  To identify novel biomarkers and gain insights to investigate phenotypic differences of MONW individuals.

SECONDARY OUTCOMES:
Postprandial profiles of lipid and inflammation | Blood will be sampled at timepoints, t = 0 minute (fasting), following the meal test, for 4 hours (t = 15, 30, 60, 90, 120, 150, 180 and 240 minutes), and pre- and post-exercise.
  Effects on fasting lipids and inflammatory markers
Measure of appetite regulation and postprandial gut hormones | Rate hunger and satiety immediately before (t=0 minute) and after meal (t=15, 30, 60, 120, 180, and 240 minutes)
  A visual analogue scale incorporating a 100-point rating scale will be used to assess each appetitive sensation, e.g. hunger, fullness, desire to eat, induced by each intervention. Gut hormones will also be measured from blood samples.
Measure of muscle and inflammation biomarkers after exercise bout | Blood samples were taken prior to the exercise and immediately after the 30-minute exercise
  Measure of muscle and inflammation biomarkers after exercise to evaluating metabolic biomarkers in energy balance
Baseline gut microbial populations and functions and relationship to the host's diet | 1 stool sample collected during study,taken at baseline (between baseline visit and before first intervention visit). Can be collected in centre or at home using a stool kit. Kit contained stabilising reagents to stabilize DNA and RNA.
  Subjects will be instructed to pass stool onto a provided dry clean stool catcher and transfer 1-5 grams stool specimen using a spatula attached to the tube lid into the stool collection leak prof tube containing preservatives.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Nutrition Research Centre, Singapore, Singapore, Singapore